CLINICAL TRIAL: NCT04127123
Title: Cloud-Based Mapping for Personalized Ablation
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty enrolling due to COVID closures
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Stanford University
Other Study IDs: 49800; 49800 (Other: Stanford IRB)
Record Dates: First submitted 2019-04-01; First posted 2019-10-15 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: arrhythmia; cardiac electrophysiology; ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation is a serious public health issue that affects over 5 million Americans in whom it may cause skipped beats, dizziness, stroke and even death. This study seeks to improve our understanding of the causes of atrial fibrillation and to design new and more effective therapy for this heart rhythm disorder.

DETAILED DESCRIPTION:
This project will focus on the development of a novel paradigm for electrophysiologic data analysis and interpretation using cloud-based computing resources and mobile technology. Currently, electrophysiologic data gathered during a procedure is analyzed by the operator using multiple separate desk-based computer systems in the electrophysiology laboratory. The investigators propose that advances in cloud-based computing resources and network connectivity should apply a mobile paradigm to apply to invasive electrophysiologic procedures.

This project will provide proof-of-concept that open-access software the investigators have developed and made available online could be used, via a mobile phone interface, to identify sites in the heart where therapy is effective. At no time will patient therapy be guided by this system. The investigators will pursue therapy using only clinical means. In parallel, a double-blinded team will analyze data in real time using our online software visualized on a smartphone. Only when the case is concluded will the data be unblinded, to determine if the mobile system was accurate in real time.

Thus, development and testing of the cloud-based computing system is designed only to establish feasibility of the paradigm, followed by improvement of computational modeling algorithms. The data that is collected will add to the investigators' existing unique catalogue of multimodal (structural, clinical, and electrophysiologic) data.

The importance of this novel paradigm is to move from analyzing large volumes of data in isolation to creating a mobile platform, and to allow scalability to increase access, such as to underdeveloped medical centers.

ELIGIBILITY:
Inclusion Criteria:

* men and women of any ethnicity
* aged 21-80 years
* undergoing ablation of atrial fibrillation at Stanford University
* failed or be intolerant of ≥ 1 anti-arrhythmic drug or not willing to accept antiarrhythmic drug therapy.

Exclusion Criteria:

* active coronary ischemia or decompensated heart failure
* atrial or ventricular clot on trans-esophageal echocardiography
* pregnancy (to minimize fluoroscopic exposure)
* inability or unwillingness to provide informed consent
* rheumatic valve disease (because it results in a unique AF phenotype)
* thrombotic disease or venous filters
* significantly reduced kidney function

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women of any ethnicity aged 21-80 years undergoing ablation at Stanford of AF. Patients will have failed or be intolerant of ≥ 1 anti-arrhythmic drug or not willing to accept antiarrhythmic drug therapy. 50 patients will be enrolled at Stanford University over 1-2 years.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Mapping Accuracy | During Procedure (Electrophysiology Study and Ablation)
  Location of driver regions for AF
Termination of atrial fibrillation | During Procedure (Electrophysiology Study and Ablation)
  Does ablation at any driver region lead to AF termination

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Narayan, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States